CLINICAL TRIAL: NCT02790762
Title: A Phase I Study of Human Umbilical Cord-Mesenchymal Stem Cells for Pneumoconiosis
Brief Title: Human Umbilical Cord-Mesenchymal Stem Cells for Pneumoconiosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Hornetcorn Bio-technology Company, LTD (Industry)
Collaborators: The Second Hospital University of South China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYK-pneumoconiosis
Record Dates: First submitted 2016-05-20; First posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Pneumoconiosis
Keywords: stem cells; Mesenchymal Stem Cells; Umbilical Cord-Mesenchymal Stem Cells; Pneumoconiosis
MeSH Terms: conditions — Pneumoconiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hUC-MSC treatment (Experimental): Patients will receive human umbilical cord mesenchymal stem cells transplantation with a 12 months follow-up.
  Interventions: Biological: Human umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Human umbilical cord mesenchymal stem cells — A single dose of 2×107 hUC-MSC will be implanted to patients by intravenous infusion, and repeated every week for four times.
  Other Names: hUC-MSC

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of human umbilical cord mesenchymal stem cell(hUC-MSC) for Pneumoconiosis.

DETAILED DESCRIPTION:
Human umbilical cord mesenchymal stem cells exhibit the potential to differentiate into mature cells typical of several tissues, which have been confirmed in in vivo and in vitro experiments.

To investigate the effects of hUC-MSC treatment for Pneumoconiosis, 10 patients with Pneumoconiosis will be enrolled and receive 4 times of hUC-MSC transplantation.

ELIGIBILITY:
Inclusion Criteria:

* The patient who have signed the informed consent document;
* Clinical and radiological evidence of liver cirrhosis.

Exclusion Criteria:

* Pregnant women or lactating mothers;
* History of neurological disease, head injury or psychiatric disorder;
* Patients with positive human immunodeficiency (HIV) at screening indicative of current of pass infection;
* With malignant tumors;
* Abnormal blood coagulation, combine other tumor or special condition;
* Patients who had participated in other clinical trials within three months prior to this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Severity of adverse events | 12 months
  According to National Cancer Institute Common Terminology Criteria for Adverse Events（NCI-CTCAE)

SECONDARY OUTCOMES:
Immunological Indicator in serum | 1, 3 ,6 and 12 months
  Expression levels of various cytokines including interferon-γ、IL-2、IL-1β、IL-4 and transforming growth factor-β1 in serum(U/ml).
The level of ceruloplasmin in serum | 1, 3 ,6 and 12 months
The level of type Ⅲ procollagen peptide in serum | 1, 3 ,6 and 12 months
Lung function as assessed by spirometry | 1, 3 ,6 and 12 months
Chest high kilovolt X-ray examination | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Guo Q Li, Professor, Principal Investigator — The second Affiliated Hospital of University of Soth China
Locations (1):
- The second Affiliated Hospital of University of Soth China, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided